CLINICAL TRIAL: NCT05921695
Title: The Relationship Between Normal Saline Infusion and Acute Kidney Injury in Patients With Heat Stroke
Brief Title: The Relationship Between Normal Saline Infusion and Acute Kidney Injury in Heat Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Yiwu Central Hospital (Other); Jinhua People's Hospital (Other); Jinhua Municipal Central Hospital (Other); Dongyang People's Hospital (Other); Lanxi People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 20230506
Record Dates: First submitted 2023-05-23; First posted 2023-06-27 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Heat Stroke
Keywords: heat stroke; normal saline; acute kidney injury; mortality
MeSH Terms: conditions — Heat Stroke; Acute Kidney Injury | interventions — Ringer's Lactate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Saline infusion group (Active Comparator): During the emergency department, the normal saline infusion was not restricted.
  Interventions: Drug: Normal Saline infusion and Ringer lactate infusion
- Ringer lactate infusion group (Experimental): Use ringer lactate or other balanced crystallographic solution instead of normal saline. Strictly limit the amount of normal saline infusion. Normal saline will only be infused by medical advice if the patient has hypochloremia or needs saline as solvent.
  Interventions: Drug: Normal Saline infusion and Ringer lactate infusion

INTERVENTIONS:
Drug: Normal Saline infusion and Ringer lactate infusion — The heat stroke patients will be infused with different chlorine concentrations fluid during the emergency department.
  Other Names: NS and Lactated Ringer's solution

SUMMARY:
The goal of this clinical trial is to compare the effect of high chlorine solution such as normal saline and non-high chlorine solution such as sodium lactate ringer's solution on renal function in patients with heat stroke. The main question it aims to answer is whether limiting the amount of normal saline infusion during emergency department can lower the incidence of acute kidney injury and mortality in patients with heat stroke.

Participants will receive a free normal saline infusion during the emergency department according to the study design, or a restricted normal saline infusion while using sodium lactate Ringer's instead.

Researchers will compare the normal saline infusion group and sodium lactate Ringer's group to see if limiting the amount of normal saline infusion during emergency department can lower the incidence of acute kidney injury and mortality in patients with heat stroke.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* diagnosed as heat stroke
* Informed consent from patients or family members.

Exclusion Criteria:

* need immediate cardiopulmonary resuscitation
* transferred from another hospital
* with original end-stage renal disease or dialysis
* with severe organ damage
* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2023-05-28 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Acute kidney injury | up to 90 days
  Acute kidney injury was defined as increase in serum creatinine by 50% within 7 days, or increase in serum creatinine by 0.3 mg/dl (26.5μmol/l) within 2 days, or oliguria

SECONDARY OUTCOMES:
Continuous renal replacement therapy | up to 90 days
  number of participants need continuous renal replacement therapy
length of ICU stay | up to 90 days
  The length patient stay in ICU
in-hospital mortality | up to 90 days
  number of participants dead in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Lan Chen, PHD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (7):
- China (7):
  - YongKang First People's Hospital, Guli, Zhejiang
  - Yiwu Central Hospital, Yiwu, Zhejiang
  - Dongyang People's Hospital, Dongyang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou
  - Jinhua Municipal Central Hospital, Jinhua
  - Jinhua People's Hospital, Jinhua
  - Lanxi People's Hospital, Lanxi